CLINICAL TRIAL: NCT01869205
Title: The Effect and Mechanism of Bronchoscopic Lung Volume Reduction by Endobronchial Valve in Korean Emphysema Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sei Won Lee, Department of Pulmonary and Critical Care Medicine and Clinical Research Center for Chronic Obstructive Airway Diseases, Asan Medical Center, University of Ulsan College of Medicine, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSCR2013-0368; A102065 (Other: Korea Healthcare Technology R&D Project)
Record Dates: First submitted 2013-06-01; First posted 2013-06-05 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Pulmonary Emphysema
Keywords: COPD; Emphysema; Bronchoscopic lung volume reduction; Endobronchial valve
MeSH Terms: conditions — Pulmonary Emphysema; Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Intervention Model Description: Bronchoscopioc lung volume reduction by endobronchial valve
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endobronchial valve: (Experimental): Endobronchial valve (size 4.0 - 7.0 mm or 5.5 - 8.5 mm) insertion for target bronchi
  Interventions: Device: Endobronchial valve

INTERVENTIONS:
Device: Endobronchial valve — One-way endobronchial valves are placed in segmental bronchi of the most hyperinflated and least perfused lobe of the emphysematous lungs on computed tomography (CT). Before the procedure, we confirm that the target lobe has no collateral ventilation with other lobes using Chartis® System (Pulmonx, Inc. Redwood City, CA, USA).
  Other Names: - EBV-TS-4.0 (Zephyr® 4.0); - EBV-TS-5.5 (Zephyr® 5.5)

SUMMARY:
To assess efficacy of bronchoscopic lung volume reduction in Korean emphysema patients

DETAILED DESCRIPTION:
The prevalence of chronic obstructive pulmonary disease (COPD) is high (13.4%). In addition, COPD ranked 10th among the causes of death in Korea, and rose to 7th in 2008. Airflow limitation of COPD is caused by a mixture of small airway disease (obstructive bronchiolitis) and parenchyma destruction (emphysema). Bronchodilator and anti-inflammatory drugs, such as corticosteroids are effective to obstructive bronchiolitis. However, these drugs are not effective to emphysema.

Lung volume reduction was devised to remove hyperinflated lung, and to function remaining lung. Surgical lung volume reduction showed improving survival in selected emphysema patients. However, surgical lung volume reduction have bee performed rarely due to significant surgery-related mortality. In this regard, non-surgical lung volume reduction methods have been developed. Of them, bronchoscopic lung volume reduction by endobronchial one-way valve is mostly used method and showed lower early complications than surgery.

The bronchoscopic lung volume reduction using endobronchial valve was proved its efficacy and safety in several large clinical trials. Although there were procedure-related complications such as acute exacerbation of COPD, pneumonia, or hemoptysis, patients receiving endobronchial valves showed improved lung functions, exercise capacity and quality of life. The endobronchial valves got approved for Conformity to European (CE) Mark in Europe. In follow-up study for patients with endobronchial valves, their efficacy and survival of patients were dependent on atelectasis induced by valves. Collateral ventilation plays a key role in endobronchial valve-induced atelectasis. Therefore, assessment of collateral ventilation should be preceded before inserting endobronchial valve.

Computed tomography (CT) can visualize and characterize morphologic change of lung of patients with COPD. Lung perfusion and ventilation CT protocols were developed for quantitative assessment of COPD before and after medical treatment. The CT protocols were expected to select optimal patients for endobronchial valves and to evaluate their efficacy.

We attempt to evaluate efficacy of bronchoscopic lung volume reduction using lung perfusion and ventilation CT and other outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 40 and below 75
* Patients with smoking history and heterogenous emphysema on chest CT
* Advanced emphysema (FEV1/FVC <70%, FEV1 of 15-45%, TLC >100% and RV >150% predicted)
* Persistent symptoms refractory to treatment
* PaCO2 <50 mmHg and PaO2 >45 mmHg
* Body mass index (BMI) ≤31.1 kg/m2 (men) or ≤32.3 kg/m2 (women)
* 6-min walk distance >140 m after pulmonary rehabilitation

Exclusion Criteria:

* Diffusing capacity (DLco) <20% predicted
* Large bullae (exceed 5 cm)
* Alpha-1 antitrypsin deficiency
* History of thoracotomy
* Excessive sputum production (throughout the week)
* Severe pulmonary hypertension ( systolic pulmonary artery pressure ≥ 45mmHg, estimated from the peak velocity of a tricuspid regurgitant jet by doppler echocardiography)
* Acute respiratory infection
* Unstable angina, congestive heart failure, or acute myocardial infarction in 6 months

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Quantitative change of lung volume on computed tomography | Before procedure and 12 weeks after procedure
  Lung perfusion and ventilation computed tomography protocols

SECONDARY OUTCOMES:
Pulmonary function test | Before procedure and 12 weeks after procedure
  Forced expiratory volume in 1s (FEV1), Forced vital capacity (FVC), Total lung capacity (TLC), Residual volume (RV)
Exercise capacity | Before procedure and 12 weeks after procedure
  Six-minute walk distance test
Healthcare quality of life | Before procedure and 12 weeks after procedure
  St. George Respiratory Questionnaire (SGRQ) and COPD Assessment Test (CAT)

CONTACTS AND LOCATIONS:
Overall Officials: Sei Won Lee, MD, Principal Investigator — Department of Pulmonary and Critical Care Medicine and Clinical Research Center for Chronic Obstructive Airway Diseases, Asan Medical Center, University of Ulsan College of Medicine, Seoul, Republic of Korea
Locations (1):
- Department of Pulmonary and Critical Care Medicine and Clinical Research Center for Chronic Obstructive Airway Diseases, Asan Medical Center, University of Ulsan College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Fishman A, Martinez F, Naunheim K, Piantadosi S, Wise R, Ries A, Weinmann G, Wood DE; National Emphysema Treatment Trial Research Group. A randomized trial comparing lung-volume-reduction surgery with medical therapy for severe emphysema. N Engl J Med. 2003 May 22;348(21):2059-73. doi: 10.1056/NEJMoa030287. Epub 2003 May 20. PMID 12759479
- [Background] Venuta F, Anile M, Diso D, Carillo C, De Giacomo T, D'Andrilli A, Fraioli F, Rendina EA, Coloni GF. Long-term follow-up after bronchoscopic lung volume reduction in patients with emphysema. Eur Respir J. 2012 May;39(5):1084-9. doi: 10.1183/09031936.00071311. Epub 2011 Oct 17. PMID 22005916
- [Background] Herth FJ, Noppen M, Valipour A, Leroy S, Vergnon JM, Ficker JH, Egan JJ, Gasparini S, Agusti C, Holmes-Higgin D, Ernst A; International VENT Study Group. Efficacy predictors of lung volume reduction with Zephyr valves in a European cohort. Eur Respir J. 2012 Jun;39(6):1334-42. doi: 10.1183/09031936.00161611. Epub 2012 Jan 26. PMID 22282552
- [Background] Hopkinson NS, Kemp SV, Toma TP, Hansell DM, Geddes DM, Shah PL, Polkey MI. Atelectasis and survival after bronchoscopic lung volume reduction for COPD. Eur Respir J. 2011 Jun;37(6):1346-51. doi: 10.1183/09031936.00100110. Epub 2010 Oct 14. PMID 20947683
- [Background] Berger RL, Decamp MM, Criner GJ, Celli BR. Lung volume reduction therapies for advanced emphysema: an update. Chest. 2010 Aug;138(2):407-17. doi: 10.1378/chest.09-1822. PMID 20682529
- [Background] Sciurba FC, Ernst A, Herth FJ, Strange C, Criner GJ, Marquette CH, Kovitz KL, Chiacchierini RP, Goldin J, McLennan G; VENT Study Research Group. A randomized study of endobronchial valves for advanced emphysema. N Engl J Med. 2010 Sep 23;363(13):1233-44. doi: 10.1056/NEJMoa0900928. PMID 20860505
- [Derived] Park TS, Hong Y, Lee JS, Oh SY, Lee SM, Kim N, Seo JB, Oh YM, Lee SD, Lee SW. Bronchoscopic lung volume reduction by endobronchial valve in advanced emphysema: the first Asian report. Int J Chron Obstruct Pulmon Dis. 2015 Jul 29;10:1501-11. doi: 10.2147/COPD.S85744. eCollection 2015. PMID 26251590